CLINICAL TRIAL: NCT06859723
Title: High Potency Cannabis: Acute and Protracted Effects
Acronym: HIGH-CAP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: California Department of Cannabis Control (DCC) (Unknown)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-5316; 93304 (Other Grant/Funding Number: CA Department of Cannabis Control)
Record Dates: First submitted 2025-02-25; First posted 2025-03-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: Abuse Cannabis; Pain; Pharmacokinetics
Keywords: THC; Cannabis
MeSH Terms: conditions — Marijuana Abuse; Pain | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Comparator: Placebo (Placebo Comparator): 0 mg THC
  Interventions: Drug: Placebo Comparator: Placebo
- Low dose THC (Active Comparator): 50 mg THC
  Interventions: Drug: Low dose THC
- High dose THC (Active Comparator): 100 mg THC
  Interventions: Drug: High dose THC

INTERVENTIONS:
Drug: Placebo Comparator: Placebo — Placebo
  Other Names: Cannabis
  Arms: Placebo Comparator: Placebo
Drug: Low dose THC — Smoked low dose THC
  Other Names: Cannabis
  Arms: Low dose THC
Drug: High dose THC — Smoked high dose THC
  Other Names: Cannabis
  Arms: High dose THC

SUMMARY:
The purpose of this research is to assess the effects of smoked cananbis when cannabis is smoked during periods of cannabis use as usual and after a brief period of abstinence.

DETAILED DESCRIPTION:
This outpatient study will assess the acute pharmacodynamic effects of smoked cannabis with ~50 mg and ~100 mg THC compared to placebo (~0 mg THC) and whether a brief period of abstinence alters these effects. Metabolism (pharmacokinetics) of THC will be examined to associate behavioral and physiological effects to plasma concentrations of THC and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* • Male or non-pregnant and non-lactating females aged 21-55 years

  * Report cannabis smoking near daily
  * Not currently seeking treatment for their cannabis use
  * Have a Body Mass Index from 18.5 - 34kg/m2.
  * Able to perform all study procedures
  * Must be using a contraceptive (hormonal or barrier methods)

Exclusion Criteria:

* Meeting DSM-V criteria for any substance use disorder other than cannabis, nicotine, caffeine
* Do not have positive urine toxicology for cannabis use during screening
* Evidence of severe psychiatric illness (e.g. mood or anxiety disorder with functional impairment or suicide risk, schizophrenia) judged by the study physician (and PI) to put the participant at greater risk of experiencing adverse events due to completion of study procedures, interfere with their ability to participate in the study, or their capacity to provide informed consent.
* Report using other illicit drugs in the prior 4 weeks
* Current predominant licit use of medical cannabis, prescription analgesics, or any medications that may affect study outcomes
* Current pain
* Pregnancy
* Currently enrolled in another research protocol
* Not using a contraceptive method (hormonal or barrier methods)
* Insensitivity to the cold water stimulus of the Cold Pressor Test
* Any disorders that might make cannabis administration hazardous as determined by evaluation physician after review of all medical assessments along with medical history.
* Not able to speak and read English

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Subject-rated drug effects of abuse liability | 3 hours
  Subject ratings of "Good Drug Effect" as measured using a visual analog scale (1-100 mm)
Analgesia as measured using the Cold Pressor Test | 3 hours
  Pain threshold assessed using the Cold Pressor Test (percent baseline)

SECONDARY OUTCOMES:
Pharmacokinetics of THC and metabolites | 3 hours
  Peak plasma levels of THC (ng/ml)
Pharmacokinetics of THC and metabolites | 3 hours
  Peak plasma levels of 11-OH-THC (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for Cannabis and Cannabinoids, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No